CLINICAL TRIAL: NCT03916328
Title: A Phase IV Open-Label Trial to Assess Bone Mineral Density in a Cohort of African Women on Depo-provera and Tenofovir Disoproxil Fumurate Switched to Tenofovir Alafenamide Fumarate Based Anti-Retroviral Therapy
Brief Title: BONE: STAR (Switching to TAF Based Anti-Retroviral Therapy) Study
Acronym: BONE:STAR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: MU-JHU CARE (Other)
Responsible Party: Principal Investigator, Flavia Kiweewa Matovu, Study Principal Investigator, MU-JHU CARE
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO-EU-380-5327
Record Dates: First submitted 2018-10-19; First posted 2019-04-16 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Bone Loss
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination; dolutegravir; Nevirapine; N,N-dimethyl-4-anisidine; Medroxyprogesterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- DMPA+ and TDF+ (Active Comparator): HIV-infected women on DMPA, and TDF containing ART.
  Interventions: Drug: TDF/3TC/EFV or DTG or NVP; Other: DMPA
- DMPA+ and B/F/TAF+ (Experimental): HIV-infected women on DMPA, and B/F/TAF.
  Interventions: Drug: B/F/TAF; Other: DMPA
- DMPA- and B/F/TAF+ (Experimental): HIV-infected women on non hormonal contraception, and B/F/TAF.
  Interventions: Drug: B/F/TAF

INTERVENTIONS:
Drug: B/F/TAF — A third of the women will be randomized to Bictergravir /Emtricitabine / Tenofovir alafenamide (B/F/TAF; Biktarvy®).
  Other Names: Biktarvy®)
  Arms: DMPA+ and B/F/TAF+; DMPA- and B/F/TAF+
Drug: TDF/3TC/EFV or DTG or NVP — A third of the women will remain on Tenofovir Disoproxil Fumurate.(TDF) containing ART.
  Arms: DMPA+ and TDF+
Other: DMPA — Two thirds of the women will be on DMPA for contraception.
  Other Names: Depo-provera
  Arms: DMPA+ and B/F/TAF+; DMPA+ and TDF+

SUMMARY:
The primarily objective of this study is to assess the effect of switching from Tenofovir Disoproxil Fumurate (TDF) to TAF based ART on bone mass and turnover among women on DMPA for contraception. HIV virologically suppressed women on DMPA will be switched from their TDF based regimen to Bictergravir /Emtricitabine / Tenofovir alafenamide (B/F/TAF; Biktarvy®) in a randomized fashion. HIV infected women on TDF and non-hormonal contraception will be switched to Biktarvy®).

ELIGIBILITY:
Inclusion Criteria:

* Age 20 through 40 years (inclusive) at screening, verified per site SOPs
* Able and willing to provide written informed consent to be screened for and to take part in the study.
* Able and willing to provide adequate locator information, as defined in site SOPs
* Previously participated in the BONE: CARE study. Additional women will be recruited from the health centers where the BONE: CARE participants were receiving HIV care, and these will be matched to those from the BONE: CARE cohort based on age, duration on ART and contraception use.
* Per participant report, plans to stay in the study catchment area in the next 24 months
* Per participant report, willing to continue using similar contraceptive method as in the BONE: CARE study.

Exclusion Criteria:

* Currently pregnant/ breastfeeding or was pregnant/ breastfeeding in the last 6 months prior to screening
* Intentions to get pregnant in the next two years
* History of active tuberculosis
* Pathologic bone fracture not related to trauma (ever)
* Has pre-existing condition known to affect bone metabolism (e.g. thyrotoxicosis, tuberculosis, diabetes mellitus, liver or renal disease)
* Is taking the following medications known to interfere with bone metabolism (steroids, anti-convulsants, bisphosphonates, cancer drugs, etc.).

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — 20 - 40 year old HIV-infected non pregnant women
Enrollment: 330 (Estimated)
Dates: Start 2019-12-03 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes in bone mineral density | 2 years
  We will assess percent change in BMD among DMPA users who switch to B/F/TAF compared to DMPA users remaining on TDF based ART
Changes in trabeculae bone score (TBS) | 2 years
  We will assess percent change in TBS among DMPA users who switch to B/F/TAF compared to DMPA users remaining on TDF based ART

SECONDARY OUTCOMES:
Changes in bone biomarkers | 2 years
  We will compare changes in bone turnover markers (CTX and P1NP) in B/F/TAF switchers with and without DMPA use

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Kiweewa Matovu, MBChB, MSc, Principal Investigator — MU-JHU CARE
Locations (1):
- MU-JHU Care Limited, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No